CLINICAL TRIAL: NCT01865071
Title: Early Closure of Temporary Loop Ileostomy After Rectal Resection for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mark Ellebaek Pedersen, Doctor, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20110026
Record Dates: First submitted 2012-10-11; First posted 2013-05-30 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Rectal Cancer
Keywords: ileostomy; rectal resection; proctectomy; stoma closure; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- loop ileostomi (Experimental): Compare early vs. late closer of the protecting ileostoma in patients requiring rectal resection for rectal cancer
  Interventions: Procedure: loop ileostomi

INTERVENTIONS:
Procedure: loop ileostomi

SUMMARY:
Early Closure of Temporary Loop Ileostomy After Rectal Resection for cancer

DETAILED DESCRIPTION:
The aim of this prospective randomized study is to compare early vs. late closer of the protecting ileostoma in patients requiring rectal resection for rectal cancer.

Early closer is defined as postoperative days 8-12 and delayed as later then 3 months.

Inclusion criteria is aged 18 years or older with rectal carcinoma, requiring rectal resection with a protecting ileostoma.

A CT-water-soluble contrast enema examination per rectum is performed at day 7, to evaluate the anastomosis in all patients. The patients will be randomized after the "intention-to-treat" principle, before the primary operation.

If there is no radiologic signs of contrast leakage ore other contraindications for early closer as septic episodes ore missing bowl movements the early closure will be preformed.

Primary end point is the rate of either postoperative death or postoperative complications occurring at 90 days after the rectal resection.

Major and minor postoperative complications (anastomotic leakage, post operative death, anastomotic fistula, postoperative peritonitis, pneumonia etc) and stoma related complications (prolapsus or peristomial eventration, erosive peristomal dermatitis, dehydration with hydroelectrolytic disorders, occlusive syndrome) would be registered.

LARS score and EORTC QLQ-30 will be sent preoperatively and after 3, 6, 12 and 24 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older.
* All patients with rectal carcinoma, requiring elective rectal resection with primary anastomosis and an protecting ileostoma
* Written informed consent was obtained from all patients

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | Death occurring during the first 90 days
  Death occurring during the first 90 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ellebæk, MD, Principal Investigator — Odense Universityhospital
Locations (1):
- Odense Universityhospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Ellebaek MB, Perdawood SK, Steenstrup S, Khalaf S, Kundal J, Moller S, Bang JC, Stovring J, Qvist N. Early versus late reversal of diverting loop ileostomy in rectal cancer surgery: a multicentre randomized controlled trial. Sci Rep. 2023 Apr 10;13(1):5818. doi: 10.1038/s41598-023-33006-4. PMID 37037856